CLINICAL TRIAL: NCT00665236
Title: Craniosacral Therapy in Migraine: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Douglas Mann, MD, Professor of Neurology, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT002750-01A2 (NIH); R21AT002750-01A2 (NIH)
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Migraine Headaches
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Craniosacral therapy administered once a week for an hour by a trained craniosacral therapist.
  Interventions: Other: Craniosacral therapy
- 2 (Active Comparator): Low-strength static magnets placed around the body for periods of up to an hour once a week.
  Interventions: Procedure: Low strength static magnets

INTERVENTIONS:
Other: Craniosacral therapy — Eight weekly 45-minute sessions with therapist
  Arms: 1
Procedure: Low strength static magnets — Placement of magnets on/around subject body by therapist; frequency: weekly for 45-minutes x 8 weeks
  Arms: 2

SUMMARY:
Treatment of migraine continues to be a major health problem today, despite many new pharmacological therapies. Limited clinical experience suggests that craniosacral therapy (CST) may be effective in the treatment of headache, including migraine. The primary aim of this proposal is to gather quality preliminary data on the usefulness of CST as an adjunct to conventional care for patients with migraine and to determine the feasibility of a larger, randomized clinical trial of CST in patients with migraine. Craniosacral therapists use a technique of gentle palpation of the head, neck and spine to release restrictions in cranial and peri-spinal tissues that are believed to contribute to a variety of health problems including headache. It is estimated that more than 2 million visits to CST practitioners are made each year, with more than 10 per cent of those for the complaint of headache. There has been no rigorous research examining the usefulness of CST for patients with migraine despite the impression of beneficial effects. Our limited preliminary data show significant, sustained benefit of CST in a small group of patients with migraine. The First Specific Aim is to determine the feasibility of developing a clinical trial comparing craniosacral therapy versus low-strength static magnets (attention-control complementary therapy) as a treatment for preventing migraine headaches. Patients with migraine, with or without aura, under care of a neurologist will be studied. After an 8-week baseline period, they will be randomized to one of two groups: 1) usual medical care plus 8 weeks of CST; or 2) usual medical care plus 8 weeks of attention-control complementary treatment. Primary outcome measures will include: 1) headache-related quality of life, 2) headache frequency, and 3) perceived benefit in those receiving treatment. The Second Specific Aim is to identify relevant secondary outcomes associated with usual care plus adjunctive craniosacral therapy for migraine. Data collection will include demographics, headache intensity and duration, health status, headache-related disability, health care utilization, and medication use. The Third Specific Aim is to identify and find solutions for potential problems in conducting a larger clinical trial to assess the efficacy of CST for the prevention of migraine. Patients will be recruited from the University of North Carolina Headache Clinic and from local neurological practices. Duration of the study for each subject is 16 weeks. Length of the entire project is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will be 12 years of age and above, either gender, meeting the 2004 International Classification of Headache Disorders (ICHD) criteria for migraine with or without aura, with a frequency of 5 to 14 per month and a headache history of more than two years. Patients must be under the care of one of the physicians participating in the study. Patients with chronic daily headache (more than 15 headache days per month) will be included only if they also have between 5 and 14 migraine headaches per month that can be clearly differentiated from chronic daily headache. Subjects or their caregivers must be willing and able to document headache characteristics and use of medications, as well as complete the assessment instruments. They must be able to come in for 8 weekly CST or LSSM interventions.

Exclusion Criteria:

* Exclusion Criteria. Patients with significant, symptomatic depression, anxiety or psychosis requiring more than two psychotropic medications daily and/or more than two visits a month to a mental health care provider; those undergoing current treatment for a major medical illness such as malignancy, autoimmune or immune deficiency disorder; pregnancy; those with clotting disorders; those with a history of head trauma or cranial or neck surgery within two years; a prior history of use of CST or magnet therapy for headache; cardiac pacemakers; other implanted or external electrical devices.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-09; Primary Completion 2009-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
HIT-6 | Post-treatment (end of 8 weeks)

SECONDARY OUTCOMES:
Headache frequency | Daily

CONTACTS AND LOCATIONS:
Overall Officials: John Douglas Mann, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Mann JD, Faurot KR, Wilkinson L, Curtis P, Coeytaux RR, Suchindran C, Gaylord SA. Craniosacral therapy for migraine: protocol development for an exploratory controlled clinical trial. BMC Complement Altern Med. 2008 Jun 9;8:28. doi: 10.1186/1472-6882-8-28. PMID 18541041
- See also: UNC's Program on Integrative Medicine — http://pim.med.unc.edu